CLINICAL TRIAL: NCT03078790
Title: Implementing a Paced Deep Breathing Module to Decrease Preoperative Anxiety in Gynecological Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Natalie A. Laska, Principle investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-005071
Record Dates: First submitted 2017-03-06; First posted 2017-03-13 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- meditation module (Experimental): The patients in this arm will be offered the meditation/deep breathing module in the pre-operative area.
  Interventions: Device: iPad

INTERVENTIONS:
Device: iPad — a 10 minute electronic guided deep breathing module offered via an iPad

SUMMARY:
Preoperative anxiety is a common occurrence for many patients undergoing all types of surgery. Patients with a high level of anxiety before surgery have been shown to have numerous negative outcomes both intra-operatively and post-operatively. Many studies have shown that preoperative psychological interventions that aim to reduce anxiety also result in improved post-operative behavioral and clinical recovery. Currently, the most common method to treat preoperative anxiety is the administration of a prescription benzodiazepine. However, there is limited clinical evidence that supports the use of sedative premedication, such as with a benzodiazepine, before surgery. Complementary integrative medical therapies including music, massage, guided imagery, and deep breathing have been proposed to minimize stress and pain in surgical patients. These therapies are thought to be effective by evoking the relaxation response through stimulation of the parasympathetic nervous system and engagement of the patient in the healing process. Relaxation and deep breathing, particularly, have been shown to reduce pain, anxiety, and "tension-anxiety" in hospitalized patients. Based on this evidence, a guided paced deep breathing module has been proposed to reduce preoperative anxiety in patients undergoing gynecological surgery at Mayo Clinic Rochester Methodist Hospital. In this study, patients' anxiety will be assessed pre-intervention on a 0-10 numeric rating scale, as well as post-intervention and a paired t-test will be used to assess effectiveness. Additionally, qualitative questions will be administered via a questionnaire post-intervention to gain more insight on the effectiveness of the intervention. The feasibility of the intervention in the busy preoperative setting will be evaluated by assessing how many times a patient is interrupted while participating in the paced deep breathing module. If this module is found to be effective in reducing patients' anxiety, it will be implemented into practice so that every patient undergoing gynecological surgery, at the institution, will be offered the module preoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Women
* aged 18 years or older
* undergoing gynecological surgery at Rochester Methodist Hospital
* roomed in pre-operative area on Eisenberg 1-4
* English-speaking
* Able to complete pre- and post-intervention questionnaires
* Able to read and understand informed consent form

Exclusion Criteria:

* Non-English speaking women
* first-case of the day gynecological surgery patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-19 (Actual)

PRIMARY OUTCOMES:
change from baseline anxiety score | recorded immediately pre-intervention and immediately post-intervention (once meditation module is complete)
  rated 0 (no anxiety) to 10 (worst anxiety possible) on a numeric rating scale

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT03078790/Prot_SAP_000.pdf